CLINICAL TRIAL: NCT04464590
Title: Interest of a Systematic One-year Monitoring by 18F-FDG PET-CT of Patients in Complete Remission of Malignant Lymphoma
Brief Title: Interest of a Systematic One-year Monitoring by 18F-FDG PET-CT
Acronym: LYMPHOTEP1
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0131
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Malignant Lymphoma; Relapsed Non Hodgkin Lymphoma; Relapsed Hodgkin's Disease, Adult; Diagnostic Imaging
Keywords: aggressive non-hodgkin lymphoma; hodgkin lymphoma; FDG-PET/CT; follow-up; routine surveillance
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the study, we aimed to characterize the role of FDG PET/CT surveillance at 12 months of malignant lymphoma in asymptomatic patients after a first complete remission and to define a rational follow-up strategy.

DETAILED DESCRIPTION:
Most aggressive lymphomas are sensitive to first-line immunochemotherapy and are in first Complete Remission (CR) with initial therapy. CR significantly decreases the risk of recurrence and increases survival. However, a cure is not guaranteed and approximately one third of lymphoma patients have a relapse disease.

FDG PET/CT is a valuable noninvasive tool in the evaluation of lymphomas, especially to differentiate viable lymphoma and fibrosis or necrosis in residual mass.

The majority of relapses are diagnosed based on clinical symptoms reported by patients. And the role of FDG PET/CT for routine surveillance of patients after treatment is controversial.

However, many medical centers use routine follow-up FDG PET/CT in addition to physical examination and laboratory analysis to detect subclinical relapse.

Thus, we can imagine a good timing to routine FDG PET/CT when the tumor burden is small in the asymptomatic window.

Survival improvement for relapse detected by routine follow-up imaging is not clearly established compared to diagnosis by clinical symptoms.

Several studies tried to assess the value of follow-up FDG PET/CT but population, type, timing and duration of surveillance imaging was very heterogeneous.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of aggressive lymphoma, complete metabolic remission after a first-line of chemotherapy, no relapse in the first year after the end of treatment

Exclusion Criteria:

* minor patient, pregnant woman, legal protection (legal curatorship / guardianship), absence of consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients were examined every 3 to 4 months during the first two years, then every 6 months for three years, including physical examination and blood-test.
  One group (group 1) of patients received a systematic routine surveillance FDG PET/CT at 12 months (PET/CT1y) according to hematologist team and the other group (group 2) did not receive routine follow-up FDG PET/CT at 12 months (non PET/CT1y).
  None patient was symptomatic the first year. A median follow-up of 24 months at the end of treatment was required.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
role of FDG-PET/CT surveillance at 12months of lymphoma in asymptomatic patient in first complete remission | one day
  detection rate of relapse at 1 year and at the end of follow-up
performances FDG-PET/CT 1 year | one day
  sensitivity, sensibility, predictive negative value, predictive positive value, accuracy

SECONDARY OUTCOMES:
overall survival and progression-free survival | one day
  as the time from the end of first-line chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: olivier delcroix, Principal Investigator — CHRU Morvan BREST Nuclear Medicine